CLINICAL TRIAL: NCT05552586
Title: The Effect of Melatonin on the Outcomes of Myocardial Ischemia/Reperfusion Injury During Coronary Artery Bypass Grafting Surgery
Brief Title: Melatonin Impact on the Outcomes of Myocardial Ischemia/Reperfusion Injury During Coronary Artery Bypass Grafting Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, eman ahmed el-said casper, Assistant lecturerer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHCL91
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Bypass Grafting; Coronary Artery Disease
Keywords: CABG; melatonin; inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Active Comparator): Melatonin Group (n=11) patients will receive 60 mg/day Melatonin capsule (M1) from the day five before surgery.
  Interventions: Dietary Supplement: Melatonin
- Control group (Placebo Comparator): Control group (n=11) patients will receive placebos with the same appearances and packaging at the same dose and time as those in the melatonin group.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — patients in the melatonin group will receive 60 mg/day Melatonin capsule (M1) from the day five before surgery.
  Arms: Melatonin group
Other: placebo — patients will receive capsules of the same size and color
  Arms: Control group

SUMMARY:
The ischemia/reperfusion (I/R) injury of the myocardium initiates a variety and complex sets of inflammatory reactions that may both exaggerate local injury as well as provoke injury of distant organ function . I/R injuries are the main causes of heart failure, morbidity, and mortality after cardiac surgery such as coronary artery bypass graft (CABG surgery) . The reactive oxygen species are believed to be excessively elevated during coronary artery bypass surgery (CABG) due to compromised free radical scavenging mechanism in the myocardium that can make myocardium highly susceptible to oxidative stress and inflammation and result in reperfusion injury .

Melatonin and its metabolites protect against inflammation by regulating several inflammatory cytokines. Additionally, melatonin is a free radical scavenger and an antioxidant agent.

the current study is designed to investigate the protective effects of melatonin against myocardial I/R injury in patients undergoing coronary artery bypass grafting (CABG) surgery.

DETAILED DESCRIPTION:
Myocardial ischemia is a situation where there is an inadequate blood and oxygen supply to the heart muscles due to partial or complete obstruction of the coronary arteries, predisposing the affected cardiac muscle to death. Hence, restoration of blood supply is critical to reestablish myocardial reperfusion. The ischemia/reperfusion (I/R) injury of the myocardium initiates a variety and complex sets of inflammatory reactions that may both exaggerate local injury as well as provoke injury of distant organ function . I/R injuries are the main causes of heart failure, morbidity, and mortality after cardiac surgery such as coronary artery bypass graft (CABG surgery) . The reactive oxygen species are believed to be excessively elevated during coronary artery bypass surgery (CABG) due to compromised free radical scavenging mechanism in the myocardium that can make myocardium highly susceptible to oxidative stress and inflammation and result in reperfusion injury . Strategies to improve the CABG related complications are much needed to augment the positive outcomes in the post-operative surviving patients. There are various therapeutic approaches to decrease or ameliorate myocardial I/R injury, these include reperfusion controlling, cardioprotective events and management via various interventions.

Melatonin (N-acetyl 5-methoxy-tryptamine) is mainly secreted by the pineal gland to regulate sleep. Since 1993 when melatonin was first reported, a wide range of melatonin functions have been directly confirmed by multiple scientific studies . Melatonin and its metabolites protect against inflammation by regulating several inflammatory cytokines. Additionally, melatonin is a free radical scavenger and an antioxidant agent. Early studies have shown that melatonin exerts beneficial effects in the context of renal I/R, myocardial I/R, and hepatic I/R. The ability to protect against I/R injury may relate to the functions of melatonin as both an anti-inflammatory and an antioxidant agent .

Some authors show an anti-apoptotic action of melatonin in different organs of the body, such as thymus, kidney, brain and liver .

the current study is designed to investigate the protective effects of melatonin against myocardial I/R injury in patients undergoing coronary artery bypass grafting (CABG) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective CABG,
* ready to participate in the study and
* can be reached by phone

Exclusion Criteria:

* • Patients who will require urgent surgery and won't have adequate time to take medications for 5 days,

  * Re-operative patients (CABG),
  * Off-pump CABG,
  * Patients who have concomitant renal failure,
  * Patients with severe respiratory problems.
  * Patients with previous stroke or significant cerebrovascular disease,
  * Patients with hepatitis b,c and HIV.
  * Inflammatory disease ex. Rheumatoid arthritis, psoriasis…,
  * Patients with ejection fraction (EF%) lower than 40%,
  * Patients undergo CABG surgery with simultaneous heart valve repair or replacement, resection of a ventricular aneurysm, or other operations.
  * Pregnancy and lactation.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Nuclear factor-kB (NF-κB) | 24 hours
  Nuclear factor-kappa B (NF-κB) is a ubiquitous transcription factor that is involved in inflammatory and immune responses, as well as in regulation of expression of many other genes related to cell survival, proliferation, and differentiation

SECONDARY OUTCOMES:
interleukin 6 il-6 | 24 hours
  Interleukin-6 is a widely used cytokine that causes inflammation and oxidative stress, which would further result in cardiac and cerebral injury. The increased expression of interleukin-6 is closely related to atherosclerosis, myocardial infarction, heart failure and ischemic stroke. It is a key risk factor for these diseases by triggering inflammatory reaction and inducing other molecules release.
Tumor necrosis factor alpha TNF-α | 24 hours
  Tumor necrosis factor (TNF) is a multifunctional cytokine that plays important roles in diverse cellular events such as cell survival, proliferation, differentiation, and death. As a pro-inflammatory cytokine, TNF is secreted by inflammatory cells, which may be involved in inflammation-associated heart diseases.
cardiac troponins | 24 hours
  cardiac marker

OTHER OUTCOMES:
LVEF% | 24 hours
  left ventricular ejection fraction
Safety (Adverse effects from melatonin) | 5 days
  Safety of melatonin
hospital length of stay | 5-7 days
  Duration of staying in hospital
ICU length of stay | 2-3 days
  Duration of staying in ICU

CONTACTS AND LOCATIONS:
Overall Officials: eman A. casper, masters, Principal Investigator — Ain shams university , faculty of pharmacy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Casper EA, Wakeel LE, Sabri NA, Khorshid R, Gamal MA, Fahmy SF. Melatonin ameliorates inflammation and improves outcomes of ischemia/reperfusion injury in patients undergoing coronary artery bypass grafting surgery: a randomized placebo-controlled study. Apoptosis. 2025 Feb;30(1-2):267-281. doi: 10.1007/s10495-024-02040-6. Epub 2024 Dec 4. PMID 39633112